CLINICAL TRIAL: NCT02585817
Title: Remote Patient Management for Cardiac Implantable Electronic Devices - A Pilot Study
Brief Title: Remote Patient Management for Cardiac Implantable Electronic Devices
Acronym: RPM-CIED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ratika Parkash (Other)
Collaborators: Cardiac Arrhythmia Network of Canada (Other); Medtronic (Industry)
Responsible Party: Sponsor-Investigator, Ratika Parkash, Staff Cardiologist, Nova Scotia Health Authority
Organization: Nova Scotia Health Authority (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RP-002
Record Dates: First submitted 2015-10-16; First posted 2015-10-23 (Estimated); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Arrhythmia, Cardiac
Keywords: Cardiac Implantable Electronic Devices
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Remote CIED Management (Experimental): Patients with a CIED will undergo remote monitoring with information technology.
  Interventions: Device: Remote CIED Management

INTERVENTIONS:
Device: Remote CIED Management — Information Technology

SUMMARY:
This is a pilot study to assess barriers, evaluate and implement a patient oriented CIED management model incorporating advanced technological innovation to promote a paradigm shift to patient-centered care involving remote CIED monitoring and programming. The advancement in technology is very important as it addresses several potential gaps and barriers in the care of patients with CIEDS:

1. Long, expensive travel for patients
2. Morbidity to patients due to delay in receiving appropriate treatment
3. Efficiency in health care delivery
4. Patient satisfaction

DETAILED DESCRIPTION:
Canada is a country with a diverse geography, of which 19% of the inhabitants are in communities classified as 'rural', but many may still have long distances to travel to reach a health care facility. This results in challenges in uniform delivery of health care throughout the country. There are 25,000 pacemaker (PM) implants and 7000 implantable defibrillator (ICD) implants yearly in Canada, with approximately 120 000 patients living with these devices. The recommended follow-up for these devices are based on consensus and position statements, with the majority of patients requiring at least yearly visits to a specialized device clinic during the lifetime of their device. During the life of these patients, many issues may arise, such as atrial or ventricular arrhythmias that may result in syncope, stroke or sudden death, need for increased monitoring resulting from device advisories, or minor programming adjustments to improve device performance, or simply the need for enhanced surveillance as the device battery depletes and replacement is anticipated.

While remote monitoring technology is currently available and has permitted surveillance and device assessment from any patient location accessible to a landline or mobile phone, the use has been inconsistent in Canada. In addition, new technology has become available that not only permits surveillance, but also remote programming of these devices. The incorporation of remote programming capability, along with automatic recalibration of device settings, allows us to develop a new paradigm of remote patient management where after the patient receives their device, they would remain in the care of their local health team and no longer require travel to the specialized 'hub' clinics for follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with an implanted pacemaker/cardiac resynchronization therapy with a pacemaker(CRT-P) capable of remote patient management would be eligible for the study that will be followed by the site where the implantation occurred OR patients with an implanted defibrillator/CRT-D capable of remote patient management where the patients reside in a community OUTSIDE of the site where the implantation occurred. The device may be de novo, existing or a patient undergoing a pulse generator change that now has remote patient management capabilities.
2. Able to provide consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Generalizability: Measurement of generalizability will be done by measuring the number of patients eligible for remote patient management as a proportion of all CIED patients. | 6 months

SECONDARY OUTCOMES:
Feasibility: Feasibility will be measured by the time to implement a fully functioning system at the participating centers | 6 months
Compliance (number of received remote transmissions divided by the number of expected remote transmissions) | 12 months
  Compliance to remote patient management will be measured for patients by the number of received remote transmissions divided by the number of expected remote transmissions.

CONTACTS AND LOCATIONS:
Overall Officials: Ratika Parkash, MD, FRCPC, Principal Investigator — Nova Scotia Health Authority
Locations (1):
- QEII HSC, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sapp JA, Gillis AM, AbdelWahab A, Nault I, Nery PB, Healey JS, Raj SR, Lockwood E, Sterns LD, Sears SF, Wells GA, Yee R, Philippon F, Tang A, Parkash R. Remote-only monitoring for patients with cardiac implantable electronic devices: a before-and-after pilot study. CMAJ Open. 2021 Jan 25;9(1):E53-E61. doi: 10.9778/cmajo.20200041. Print 2021 Jan-Mar. PMID 33495385